CLINICAL TRIAL: NCT06959537
Title: A Phase Ib Study of Novel Combination (New) of Low Dose Oral CyclophoSphamide (s) to Potentiate Axatilimab (A) + Retifanlimab (R) in Treating Metastatic Triple Negative Breast Cancer (TNBC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0016; NCI-2025-03170 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; axatilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Cyclophosphamide + Axatilimab + Retifanlimab (Experimental): Participants will be requestd to maintain a medication diary of each dose of medication while taking oral cyclophosphamide. The medication diary will be returned to clinic staff at the end of each course.
  Interventions: Drug: Cyclophosphamide; Drug: Axatilimab (SNDX-6352); Drug: Retifanlimab

INTERVENTIONS:
Drug: Cyclophosphamide — Given by mouth
Drug: Axatilimab (SNDX-6352) — Given by IV
Drug: Retifanlimab — Given by IV

SUMMARY:
The goal of this clinical research study is to find the best dose of the drugs cyclophosphamide and axatilimab that can be given in combination with the standard dose of retifanlimab to patients with metastatic TNBC.

DETAILED DESCRIPTION:
Primary Objective:

The goal of this clinical research study is to find the best dose of the drugs cyclophosphamide and axatilimab that can be given in combination with the standard dose of retifanlimab to patients with metastatic TNBC.

Secondary Objectives:

The goal of this clinical research study is to find the best dose of the drugs cyclophosphamide and axatilimab that can be given in combination with the standard dose of retifanlimab to patients with metastatic TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or locally recurrent unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients must have histologically or cytologically confirmed non-IBC triple negative breast cancers, defined here as ER<1%, PR<1% and HER2 negative per ASCO CAP 2018 guideline. OR
* Inflammatory breast cancer (IBC) confirmed according to international consensus criteria that is ER<20% and PR<20%.
* At least 1 week since prior chemotherapy or radiation therapy
* Age .18 years.
* Has at least one measurable lesion per RECIST 1.1
* ECOG performance status . 2 (Karnofsky . 60%,).
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count . 1,000/mcL
  * hemoglobin >9 mg/dL
  * platelets . 100,000/mcL
  * total bilirubin . institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) . 3 ~ institutional ULN; . 5 ~ institutional ULN if confirmed liver metastasis and elevation is deemed to be directly due to metastasis.
  * Creatinine clearance .30 mL/min (measured by the Cockcroft-Gault equation*).
* Ability to understand and the willingness to sign a written informed consent
* . Cognitively impaired subjects will not be enrolled in this study.
* Negative serum pregnancy test within 72 hours of receiving the first dose of the study medication for women of childbearing potential as per institutional guidelines.
* Subjects of childbearing potential must be willing to use highly effective birth control methods or be surgically sterile or abstain from heterosexual activity for the course of the study. Women must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.

    * Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
    * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of all study drug administration.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) except for alopecia. Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to > Grade 2 for at least 3 months prior to [enrollment/Cycle 1 Day 1] and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, including: Chemotherapyinduced neuropathy, Fatigue, Residual toxicities from prior IO treatment: Grade 1 or Grade 2 endocrinopathies which may include: Hypothyroidism/hyperthyroidism, Type I diabetes, Hyperglycemia, Adrenal insufficiency, Adrenalitis and Skin hypopigmentation (vitiligo)
* Patients with a history of interstitial lung disease (past or current) or active, non-infectious pneumonitis.
* Patients with active autoimmune disease requiring systemic immunosuppression with corticosteroids (> 10 mg/day of prednisone or equivalent) or immunosuppressive drugs within 2 years before the first dose of study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide, axatilimab, retifanlimab used in study.
* Patients with uncontrolled intercurrent illness. Medical history or complication considered inappropriate for participation in the study, or a serious physical or psychiatric disease, the risk of which may be increased by participation in the study in the investigator's opinion.
* Patients with active infections requiring systemic antibiotics or antifungal or antiviral treatment within 14 days of C1D1 study treatment.
* Patients with known active Hepatitis B or Hepatitis C infection. Testing is required to establish eligibility. Active Hepatitis B infection is defined as a positive Hepatitis B surface antigen and positive Hepatitis B core antibody test. Active Hepatitis C infection is defined assay.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured.

For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

* Patients with known HIV infection, defined as positive for HIV1/2 antibodies. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study due to potential for teratogenic or abortifacient effects.
* Patients who are cancer survivors other than cured non-melanomatous skin cancer or cured cervical carcinoma in situ and thyroid cancer will be excluded from the study as other cancers can recur.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with active brain metastasis if treatment is warranted. Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)- directed therapy shows no evidence of progression.
* Patients with known leptomeningeal disease, defined as unequivocal imaging or cytologyproven disease.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better, and EF greater than 45% despite best supportive cae.
* Patients with a history or presence of screening ECG test that is clinically significantly abnormal in the investigator's opinion. Patients with a prolonged Qtc interval > 480 milliseconds (corrected by Fridericia or Bazett formula are excluded, but medically controlled arrhythmias are allowed.
* Patients with a history of significant cardiac event within 6 months of C1D1. Significant cardiac events include baseline NYHA class III/IV cardiac disease, acute myocardial infarction, severe/unstable angina, cardiomyopathy, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, critical conduction delay, transient ischemic attack or pulmonary embolism.
* Patients who are receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Bora Lim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org